CLINICAL TRIAL: NCT03103217
Title: Exploring the Effectiveness of a Brief CBT Intervention for Anxious Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC 16012
Record Dates: First submitted 2016-03-21; First posted 2017-04-06 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Brief CBT intervention (Experimental)
  Interventions: Behavioral: brief CBT for anxious pregnant women

INTERVENTIONS:
Behavioral: brief CBT for anxious pregnant women — one off 3 hour session including psychoeducation, exploration of cognitions and experiential practice of behavioural techniques.

SUMMARY:
Pregnancy is a time of significant adjustment and uncertainty. Anxiety is common among this group and is associated with poor cognitive and physical outcomes for both the mother and child. Few trials have been conducted to ascertain the effectiveness of brief psychological interventions designed to alleviate general anxiety, labour and pregnancy specific anxiety and promote well being.

The aim of this project is to establish if a brief Cognitive Behavioural Therapy treatment is effective in reducing general anxiety during pregnancy. The study will also explore whether the treatment has an impact on reducing pregnancy specific and labour related anxiety and reducing medical intervention.

DETAILED DESCRIPTION:
This study is a prospective matched cohort design with follow up. The treatment group will consist of women who attend once to a one off 3 hour brief cognitive behavioural therapy treatment (CBT) session. Outcome measures will be completed at 3 time points, baseline, 2 weeks post intervention and 2 weeks' post partum (follow up).

A previously published dataset collected locally will be used as a control group. This dataset includes 120 sets of data who have completed the Hospital Anxiety and Depression Scale (HADS) which will be the primary outcome measure for this study. Furthermore, the dataset includes data on several key variables including age, current pregnancy information, past pregnancy information, family and partner support available, medical support/input, income, education, living circumstances and future plan. These will be matched at key variables which are predictors of anxiety during pregnancy and might otherwise be expected to influence scores on outcome variables and utilised as covariates. The outcome measures will be completed at the same time points follow up, 2 months' post partum.

As part of a preexisting maternity care system, women are routinely offered a stress reduction session by their community midwives. Those who wish to attend are routinely placed on a database. For the purpose of this research, everyone who has been put forward for the group will be sent a covering letter, personal Information sheet (PIS) and screening HADS by the lead clinician (Mo Tabib - midwife). Participants who express an interest will be invited to have a telephone consultation with the chief Investigator. During this telephone call, eligibility will be discussed ad if appropriate telephone consent will be sought. Following this, those who do not meet eligibility criteria will be invited to attend the session as planned at Aberdeen Maternity Hospital and continue with their maternity care as usual. Eligible participants will be sent a pack of baseline measures as well as a consent form. Participants will have the option of returning these in a pre paid envelope or deposit in a confidential box at the session. Consent will also be sought for access to online medical records and consent to contact participants following the group by phone/text/email as reminder. Participants will be emailed two weeks following the session as a reminder to complete second set of measures. Participants will identify three areas which they will commit to practice following the session. The chief investigator will track their delivery date using using an online care system; 2 months' post-partum they will receive a further reminder text to complete final questionnaire set.

The chief researcher will seek informed, telephone consent initially, which can be withdrawn at any time. Consent will be discussed with potential participants during a telephone consultation following being sent the PIS and screening tool. If potential participants are interested and eligible the chief researcher will send out a consent form by means of written consent where participants will be offered choice of returning in post or deposit in a confidential box at the session. It will be highlighted that participants can withdraw from the study at any point.

ELIGIBILITY:
Inclusion Criteria:

* - Pregnant woman
* Referred to group and screened for suitability
* Attended brief pregnancy session
* Contact with community midwife
* General anxiety (Score >8 on HADS)
* Able to read, write and understand English
* Aged over 16
* Ability to give consent

Exclusion Criteria:

* Exclusion criteria will include severe mental health problems such as severe depression with suicidal ideation, psychosis, personality disorder; terminal illness; inability to give informed consent in English, and inability to understand written and spoken English as questionnaires are not standardized in other languages.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to post intervention and at follow-up -Hospital depression and anxiety scale | baseline, 2 weeks and 2 months

SECONDARY OUTCOMES:
Change from Baseline to post intervention - Pregnancy Related Anxiety Questionnaire - Short | baseline and 2 weeks
Change from Baseline to post intervention and at follow-up - The Warick Edinburgh Mental Well-being scale | baseline, 2 weeks and 2 months
Childbirth experience questionnaire | 2 months only

CONTACTS AND LOCATIONS:
Overall Officials: Paul Morris, Health Psychology, Study Chair — University of Edinburgh
Locations (1):
- Victoria Ross, Aberdeen, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No